CLINICAL TRIAL: NCT00002363
Title: Study of the Safety and Effects of Two Doses of SPC3, Administered Daily Intravenously in HIV-1 Seropositive Patients
Brief Title: The Safety and Effectiveness of SPC3 in HIV-1 Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia Research Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 257A; SPC3-US1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Metabolism

INTERVENTIONS:
Drug: Peptide Construction 3, Synthetic

SUMMARY:
To assess the effects of two doses of synthetic peptide construction 3 ( SPC3 ) on HIV-1 plasma levels (as measured by RNA PCR Amplicor) and on lymphocyte subsets in patients with initial viral load above 10,000 copies/ml. To study the safety of SPC3 and the kinetics of HIV-1 plasma level changes.

DETAILED DESCRIPTION:
The first five patients receive SPC3 daily for 3 weeks. If that dose is tolerated, the dose is increased and given to the next 5 patients for 3 weeks. The remaining ten patients receive a dose of SPC3 based on response to the previous two dose levels. Patients are followed through day 28.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretrovirals provided regimen has been stable for at least 6 weeks prior to study screening.

Patients must have:

* HIV seropositivity for at least 6 months.
* CD4 >= 100 cells/mm3.
* HIV RNA PCR (Amplicor) > 10,000 copies/ml.
* No significant active opportunistic infection or tumor at study entry.

FDA DISCLAIMER:

* The FDA encourages the inclusion of females of childbearing potential in study protocols, but the sponsor of this protocol specifically excludes females of childbearing potential from this study and includes only females who are sterile. Any questions about these inclusion/exclusion criteria should be directed to the study's contact person.

Prior Medication:

Allowed:

* Prior antiretrovirals.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

Inability to communicate with investigator or deemed likely to be noncompliant on study.

Concurrent Medication:

Excluded:

* Any drug that may interact with SPC3 (e.g., suramin).

Patients with the following prior condition are excluded:

History of relevant drug hypersensitivity.

Prior Medication:

Excluded:

* Investigational drug within the past 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (1):
- Brown Univ School of Medicine, Providence, Rhode Island, United States